CLINICAL TRIAL: NCT06752083
Title: Evaluation of the Efficacy and Safety of an AHCC®-Based Supplement (Lentinula Edodes) in Promoting Negativity of Persistent HPV Infection: A Retrospective Multicenter Clinical Study
Brief Title: Efficacy of Lentinula Edodes-Derived Supplement (AHCC®) in Promoting Negativity of Persistent HPV Infection
Status: Completed | Type: Observational
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Other Study IDs: 117_22.112024_Papion®
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Active Hexose Correlated Compound; Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unvaccinated with AHCC® Supplement: Women previously managed in routine clinical practice with AHCC® supplementation alone for persistent HPV infection. Participants had not received HPV vaccination prior to treatment. Clinical data were retrospectively collected from medical records to evaluate HPV-DNA clearance following this real-world management strategy.
  Interventions: Dietary Supplement: AHCC® (Active Hexose Correlated Compound)
- Vaccinated with AHCC® Supplement: Women previously managed in routine clinical practice with combined AHCC® supplementation and nonavalent HPV vaccination for persistent HPV infection. Treatments were prescribed as part of standard care. Clinical data were retrospectively collected to assess HPV-DNA clearance following combined real-world exposure.
  Interventions: Dietary Supplement: AHCC® (Active Hexose Correlated Compound); Biological: Gardasil 9®
- Vaccinated Only: Women previously managed in routine clinical practice with nonavalent HPV vaccination alone for persistent HPV infection. No AHCC® supplementation was used. Clinical data were retrospectively collected to assess HPV-DNA clearance following vaccination as standard care.
  Interventions: Biological: Gardasil 9®

INTERVENTIONS:
Dietary Supplement: AHCC® (Active Hexose Correlated Compound) — AHCC® supplementation previously prescribed as part of routine clinical care. Information on dosage and duration was retrospectively collected from medical records.
  Other Names: Lentinula edodes supplement, Papion®
  Groups: Unvaccinated with AHCC® Supplement; Vaccinated with AHCC® Supplement
Biological: Gardasil 9® — Nonavalent HPV vaccination previously administered as part of routine clinical care. Vaccination status was retrospectively obtained from medical records.
  Groups: Vaccinated Only; Vaccinated with AHCC® Supplement

SUMMARY:
This is a retrospective, multicenter, observational study evaluating real-world HPV-DNA clearance in women with documented persistent high-risk HPV infection lasting at least six months. Clinical data were retrospectively collected from medical records of women managed in routine practice with one of three strategies: AHCC® supplementation alone, nonavalent HPV vaccination alone, or the combination of AHCC® supplementation and nonavalent HPV vaccination. The primary objective is to assess HPV-DNA clearance at 4 and 6 months following treatment initiation.

DETAILED DESCRIPTION:
This retrospective, multicenter, observational study evaluates HPV-DNA clearance in women with documented persistent high-risk HPV infection managed in routine clinical practice. Eligible participants had confirmed HPV-DNA positivity persisting for at least six months and no high-grade cervical lesions.

Clinical data were retrospectively collected from medical records from January 2023 to December 2024. Participants were categorized into three exposure groups based on treatments already received as part of standard care: AHCC® supplementation alone, nonavalent HPV vaccination alone, or combined AHCC® supplementation and nonavalent HPV vaccination. No randomization or prospective treatment assignment was performed.

The primary outcome is HPV-DNA clearance, defined as conversion from HPV-DNA positive to negative status, assessed at 4 and 6 months after treatment initiation. Secondary outcomes include safety, tolerability, and treatment compliance based on routinely collected clinical data. This study reflects real-world clinical practice and was not designed as a randomized interventional trial.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 years or older.
* Documented persistent high-risk HPV infection for at least 6 continuous months, confirmed by consecutive HPV-DNA tests.
* Absence of high-grade cervical lesions (≤ CIN1).
* Availability of complete clinical records with evaluable HPV-DNA testing at baseline and follow-up.
* Documented management with AHCC® supplementation alone, nonavalent HPV vaccination alone, or combined AHCC® supplementation and nonavalent HPV vaccination in routine clinical practice.
* No prior excisional or ablative treatment of the cervix (including conization or LEEP).

Exclusion Criteria:

* History of cervical excisional or ablative treatment (including conization or LEEP).
* Presence of high-grade cervical lesions (CIN2 or worse) or invasive cervical cancer.
* Incomplete clinical documentation or missing HPV follow-up data.
* Conditions known to significantly alter immune function, including ongoing immunosuppressive therapy, active autoimmune disease requiring systemic treatment, or documented immunodeficiency, when such information was available in medical records.
* Prior systemic antiviral or immunomodulatory therapy specifically aimed at HPV clearance during the observation period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This retrospective study includes only female patients because cervical HPV infection and related clinical outcomes are specific to female reproductive anatomy. Sex was determined from routinely collected medical record data.
Study Population: Women with documented persistent high-risk HPV infection for at least six months whose clinical data were retrospectively identified from medical records at multiple participating gynecology centers.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
HPV-DNA Clearance Rate | 4 months and 6 months
  Proportion of participants achieving HPV-DNA negativity, defined as conversion from HPV-DNA positive to negative status based on clinically validated HPV-DNA testing.

SECONDARY OUTCOMES:
Safety and Tolerability | 4 months and 6 months
  Description of adverse events, tolerability, and treatment compliance based on retrospective review of routinely collected clinical records. Adverse events were classified according to CTCAE version 5.0 and analyzed descriptively.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gau VL, Benninger MS. Potential Role for Active Hexose Correlated Compound (AHCC) in Treatment of Recurrent Respiratory Papillomatosis. J Voice. 2022 Jul;36(4):441-442. doi: 10.1016/j.jvoice.2022.05.004. Epub 2022 Jun 27. No abstract available. PMID 35773058
- [Background] Smith JA, Mathew L, Gaikwad A, Rech B, Burney MN, Faro JP, Lucci JA 3rd, Bai Y, Olsen RJ, Byrd TT. From Bench to Bedside: Evaluation of AHCC Supplementation to Modulate the Host Immunity to Clear High-Risk Human Papillomavirus Infections. Front Oncol. 2019 Mar 20;9:173. doi: 10.3389/fonc.2019.00173. eCollection 2019. PMID 30949451
- [Background] Smith JA, Gaikwad AA, Mathew L, Rech B, Faro JP, Lucci JA 3rd, Bai Y, Olsen RJ, Byrd TT. AHCC(R) Supplementation to Support Immune Function to Clear Persistent Human Papillomavirus Infections. Front Oncol. 2022 Jun 22;12:881902. doi: 10.3389/fonc.2022.881902. eCollection 2022. PMID 35814366